CLINICAL TRIAL: NCT07037537
Title: To Evaluate the Efficacy and Safety of Laparoscopic-assisted Nipple-areola-sparing Mastectomy Plus Pectoral Anterior Prosthesis Plus Mesh Immediate One-step Breast Reconstruction Plus Concurrent Autologous Fat Grafting: a Prospective, Single-centre, Single-arm Study
Brief Title: Evaluation of the Effectiveness and Safety of Laparoscopic Assisted Mastectomy With Preservation of Nipple and Areola, Immediate One-step Breast Reconstruction With Pectoral Muscle Prosthesis and Patch, and Simultaneous Autologous Fat Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-362
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Patients
Keywords: Breast cancer; Endoscopic technology; Breast reconstruction surgery; Autologous fat transplantation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic assisted NSM+breast reconstruction+simultaneous fat transplantation (Experimental): Endoscopic assisted NSM+prosthesis combined with patch for anterior breast reconstruction and simultaneous fat transplantation
  Interventions: Procedure: Endoscopic assisted NSM+breast reconstruction+simultaneous fat transplantation

INTERVENTIONS:
Procedure: Endoscopic assisted NSM+breast reconstruction+simultaneous fat transplantation — Laparoscopic assisted mastectomy with preservation of nipple and areola, combined with chest muscle anterior prosthesis and patch, immediate one-step breast reconstruction and simultaneous autologous fat transplantation

SUMMARY:
Evaluation of the effectiveness and safety of laparoscopic assisted breast resection with preservation of nipple and areola, combined with chest muscle anterior prosthesis and patch for immediate one-step breast reconstruction and concurrent autologous fat transplantation in a prospective study

DETAILED DESCRIPTION:
This study is a prospective, single center, single arm clinical trial. It is planned to recruit 29 patients with unilateral breast cancer of cT1-2N0M0. Patients who meet the inclusion criteria are planned to undergo laparoscopic assisted NSM+prosthesis combined with patch breast reconstruction and concurrent fat transplantation surgery.

Main endpoint of the study: incidence of severe complications after breast reconstruction surgery.

Secondary study endpoints: BREAST-Q (Breast Reconstruction Module) score, breast reconstruction success rate, incidence of all complications, physician evaluated breast cosmetic outcomes, occurrence of capsule contractures, nipple areola and breast skin sensation, and tumor safety.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 70 years old;
2. In the first diagnosis of unilateral breast cancer patients, the maximum diameter of invasive tumor is ≤ 5cm, and there is no requirement for tumor size of carcinoma in situ in principle;
3. Patients undergoing preventive mastectomy are not allowed to be included in the study;
4. Clinical examination and auxiliary examinations suggest that the tumor is confined to the mammary gland and has not invaded the nipple areola complex, skin, or chest wall;
5. Clinical axillary lymph node negative (clinical physical examination and imaging suggest negative axillary lymph nodes; for suspected positive axillary lymph nodes, fine needle aspiration or hollow needle biopsy is required to confirm negative);
6. Sentinel lymph node biopsy negative;
7. Patients with low load positive axillary lymph nodes (isolated tumor cells, micro or macro metastases), but exempted from adjuvant radiotherapy after surgery;
8. Patients who are not suitable for breast conserving surgery or who are unwilling to undergo breast conserving surgery and plan to undergo laparoscopic assisted mastectomy with preservation of the nipple and areola, as well as immediate one-step breast reconstruction with a breast prosthesis combined with a chest muscle prosthesis and simultaneous fat transplantation; If frozen pathology or routine pathology indicates a positive posterior margin of the nipple, it is allowed to remove the nipple, but the areola must be preserved;
9. The volume of the prosthesis is less than 500cc;
10. During the observation period of the study, the affected side may consider re fat injection, but symmetrical surgery is not allowed on the healthy side;
11. ECOG score 0-1 points;
12. New adjuvant chemotherapy patients are allowed to be enrolled;
13. No smoking history or quitting smoking for at least 4 weeks;
14. The researcher determines that they are able to comply with the research protocol;
15. Those who participate in other clinical trials (including intervention or non intervention studies) at the same time and are judged by the researchers to not affect the study protocol can be enrolled normally;
16. After obtaining sufficient information, voluntarily participate and sign an informed consent form.

Exclusion Criteria:

1. Specialized physical examination and/or auxiliary examination suggest that the tumor involves the nipple areola complex (including Paget's disease) or the skin;
2. Double breast cancer;
3. Bilateral breast reconstruction patients;
4. Patients who have undergone fat injection, breast augmentation with implants, and breast reduction surgery in the past;
5. Patients with incomplete immune function, poor control of diabetes and active smoking;
6. Patients with severe breast sagging;
7. Breast cup size ≥ E;
8. Accept two-step breast reconstruction using dilators/prostheses, autologous breast reconstruction, and breast reconstruction performed through open surgery;
9. Patients who have previously received and/or received postoperative radiotherapy for the reconstruction site or chest wall;
10. Patients who plan to undergo symmetrical surgery on the healthy breast during the visit period;
11. Patients with mental illnesses or abnormalities who are expected to be unable to independently complete the BREAST-Q scale;
12. Pregnant and lactating patients;
13. Poor compliance, unable to conduct relevant examinations and follow ups according to the trial requirements;
14. Suffering from serious accompanying diseases or other comorbidities that may interfere with planned treatment, or any other circumstances that the researcher deems unsuitable for the patient to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious complications after breast reconstruction surgery | One week after surgery, one month after surgery, three months after surgery, six months after surgery, and one year after surgery
  All surgical related complications (including hematoma, poor wound healing, skin flap necrosis, infection, incision dehiscence, fat injection related complications, etc.) are classified according to the Clavien Dindo scoring system. The Clavien Dindo grading system is based on the severity of postoperative complications and whether corresponding treatment is needed for the complications. Postoperative complications are classified into grades I-V, and those classified as grade III or above by Clavien Dindo are considered serious complications.

SECONDARY OUTCOMES:
BREAST-Q (Breast Reconstruction Module) score | BREAST-Q scoring was performed at preoperative, postoperative 1-month, 3-month, 6-month, and 12-month follow-up
  This experiment obtained subject report results from four dimensions of breast satisfaction, psychological health, physical health, and sexual health using the BREAST-Q (Breast Reconstruction Module) scoring system. BREAST-Q scoring was performed at preoperative, 1 month, 3 months, 6 months, and 12-month follow-up. The BREAST-Q score at 12 months after surgery is the main evaluation metric.
Success rate of breast reconstruction | One year after surgery
  Calculation formula:The result of subtracting the number of implant removal cases caused by complications from the total number of breast reconstruction cases received, divided by the total number of reconstruction cases received.Definition of implant removal caused by complications: Refers to the removal of implants during the 12-month follow-up period due to surgical related reasons such as hematoma, serum swelling, skin flap necrosis, nipple areola necrosis, infection, incision dehiscence, implant exposure, capsule contraction, and prosthesis displacement.
All incidence of complications | On the day of surgery, one week after surgery, one month after surgery, three months after surgery, six months after surgery, and one year after surgery
  Complications such as hematoma, poor wound healing, skin flap necrosis, infection, incision dehiscence, and fat injection related complications are classified according to the Clavien Dindo scoring system, including grades I-V, and evaluated and recorded.
Breast cosmetic effects evaluated by doctors | Before surgery，on the day of surgery, one months after surgery,three months after surgery, six months after surgery, and one year after surgery
  The cosmetic effect of breast reconstruction is evaluated by professional doctors independent of the surgeon using the ueda scoring criteria based on patient photos.
Occurrence of capsule contraction | one months after surgery,three months after surgery, six months after surgery, and one year after surgery
  The Baker classification method (Spear&Baker, 1995) was used for evaluation.
Nipple, areola, and breast skin sensation | Before surgery, one week after surgery, one months after surgery,three months after surgery, six months after surgery, and one year after surgery
  The Semmes Weinstein single filament inspection method was used to measure tactile sensation. Semmes Weinstein Monofilament Inspection Method
Tumor safety | five years after surgery
  Disease free survival (DFS) and overall survival (OS). DFS defines the time from surgery to the occurrence of recurrence, metastasis, or last follow-up. OS defines the time from surgery to patient death or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: xiuchun chen, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Result] Kraenzlin F, Chopra K, Kokosis G, Venturi ML, Mesbahi A, Nahabedian MY. Revision Breast Reconstruction with Prepectoral Pocket Conversion of Submuscular Breast Implants. Plast Reconstr Surg. 2021 May 1;147(5):743e-748e. doi: 10.1097/PRS.0000000000007885. PMID 33890886
- [Result] Chatterjee A, Nahabedian MY, Gabriel A, Macarios D, Parekh M, Wang F, Griffin L, Sigalove S. Early assessment of post-surgical outcomes with pre-pectoral breast reconstruction: A literature review and meta-analysis. J Surg Oncol. 2018 May;117(6):1119-1130. doi: 10.1002/jso.24938. Epub 2018 Jan 18. PMID 29346711
- [Result] Li Y, Xu G, Yu N, Huang J, Long X. Prepectoral Versus Subpectoral Implant-Based Breast Reconstruction: A Meta-analysis. Ann Plast Surg. 2020 Oct;85(4):437-447. doi: 10.1097/SAP.0000000000002190. PMID 31913902
- [Result] Feng Y, Liang F, Wen N, Yang H, Zhou J, Zhang S, Liu X, Qiu M, Xie Y, Du Z. An Innovative and Highly Efficient Single-Port Endoscopic Nipple-/Skin-Sparing Mastectomy and Dual-Plane Direct-to-Implant Breast Reconstruction: A Prospective Study from a Single Institution. Aesthetic Plast Surg. 2024 Mar;48(6):1133-1141. doi: 10.1007/s00266-023-03402-2. Epub 2023 May 30. PMID 37253841
- [Result] Mok CW, Lai HW. Endoscopic-assisted surgery in the management of breast cancer: 20 years review of trend, techniques and outcomes. Breast. 2019 Aug;46:144-156. doi: 10.1016/j.breast.2019.05.013. Epub 2019 May 20. PMID 31176887
- [Result] Wang ZH, Gao GX, Liu WH, Wu SS, Xie F, Xu W, Ding GQ, Xu YQ, Zhang ZT, Qu X. Single-port nipple-sparing subcutaneous mastectomy with immediate prosthetic breast reconstruction for breast cancer. Surg Endosc. 2023 May;37(5):3842-3851. doi: 10.1007/s00464-023-09862-6. Epub 2023 Jan 25. PMID 36695902
- [Result] Li L, Su Y, Xiu B, Huang X, Chi W, Hou J, Zhang Y, Tian J, Wang J, Wu J. Comparison of prepectoral and subpectoral breast reconstruction after mastectomies: A systematic review and meta analysis. Eur J Surg Oncol. 2019 Sep;45(9):1542-1550. doi: 10.1016/j.ejso.2019.05.015. Epub 2019 May 14. PMID 31256950
- [Result] Abbate O, Rosado N, Sobti N, Vieira BL, Liao EC. Meta-analysis of prepectoral implant-based breast reconstruction: guide to patient selection and current outcomes. Breast Cancer Res Treat. 2020 Aug;182(3):543-554. doi: 10.1007/s10549-020-05722-2. Epub 2020 Jun 9. PMID 32514624
- [Result] Ostapenko E, Nixdorf L, Devyatko Y, Exner R, Wimmer K, Fitzal F. Prepectoral Versus Subpectoral Implant-Based Breast Reconstruction: A Systemic Review and Meta-analysis. Ann Surg Oncol. 2023 Jan;30(1):126-136. doi: 10.1245/s10434-022-12567-0. Epub 2022 Oct 16. PMID 36245049
- [Result] Rancati AO, Angrigiani CH, Hammond DC, Nava MB, Gonzalez EG, Dorr JC, Gercovich GF, Rocco N, Rostagno RL. Direct to Implant Reconstruction in Nipple Sparing Mastectomy: Patient Selection by Preoperative Digital Mammogram. Plast Reconstr Surg Glob Open. 2017 Jun 20;5(6):e1369. doi: 10.1097/GOX.0000000000001369. eCollection 2017 Jun. PMID 28740781
- [Result] Sigalove S. Prepectoral breast reconstruction and radiotherapy-a closer look. Gland Surg. 2019 Feb;8(1):67-74. doi: 10.21037/gs.2019.01.01. PMID 30842930
- [Result] Sorrentino L, Regolo L, Scoccia E, Petrolo G, Bossi D, Albasini S, Caruso A, Vanna R, Morasso C, Mazzucchelli S, Truffi M, Corsi F. Autologous fat transfer after breast cancer surgery: An exact-matching study on the long-term oncological safety. Eur J Surg Oncol. 2019 Oct;45(10):1827-1834. doi: 10.1016/j.ejso.2019.05.013. Epub 2019 May 21. PMID 31133371
- [Result] Gronovich Y, Winder G, Maisel-Lotan A, Lysy I, Sela E, Spiegel G, Carmon M, Hadar T, Elami A, Eizenman N, Binenboym R. Hybrid Prepectoral Direct-to-Implant and Autologous Fat Graft Simultaneously in Immediate Breast Reconstruction: A Single Surgeon's Experience with 25 Breasts in 15 Consecutive Cases. Plast Reconstr Surg. 2022 Mar 1;149(3):386e-391e. doi: 10.1097/PRS.0000000000008879. PMID 35196670